CLINICAL TRIAL: NCT03980639
Title: Abatacept and the Risk of Cancer: a Case Non-case Analysis in VigiBase
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0440
Record Dates: First submitted 2019-01-18; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Antirheumatic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- abatacept: patients with abatacept prescription
  Interventions: Drug: patient treated with DMARD
- others bDMARDs: patients with at least one bDMARD prescriptions
  Interventions: Drug: patient treated with DMARD

INTERVENTIONS:
Drug: patient treated with DMARD — Case report of cancer overall

SUMMARY:
There are very few data on the safety of Biologic Disease Modifying Anti-Rheumatic Drugs (bDMARDs), especially abatacept which compared to Tumor Necrosis Factor α (TNFα) inhibitors has distinct mechanism of action. Abatacept is a recombinant fusion protein of human Cytotoxic T-Lymphocyte Antigen 4 (CTLA-4) and the Fc region of human immunoglobulin gamma-1 (IgG1). This CTLA4-fusion protein blocks the signal of T cell activation by binding to CD80 and CD86.

Recently, the investigator's study found in a US cohort of 64,000 patients with Rheumatoid Arthritis (RA) a potential signal for a higher risk of cancer overall and particularly non-melanoma skin cancer with abatacept compared to other bDMARDs (article in press). These results were in accordance with another prospective cohort study of the public health care system in Sweden, showing an increased risk of NMSC in abatacept users compared with TNFα inhibitors. As these results warrant replication, the present study will assess whether abatacept is associated with an increased risk of reporting overall cancer and specific cancer, including breast, lung, lymphoma, cervical, melanoma and NMSC, compared to other bDMARDs.

DETAILED DESCRIPTION:
A case non-case study using Vigibase®, the World Health Organization Global Individual Case Safety Reports (ICSRs) database which includes more than 18 million reports forwarded to the WHO Uppsala Monitoring Center by national pharmacovigilance systems from over 130 countries around the world since 1967. Information on the adverse effects reported include patient demographics and medical relevant history, drugs recorded according to the WHO Drug dictionary and adverse drug reactions coded with Medical Dictionary for Regulatory Activities (MedDRA) terms will be perform.

ELIGIBILITY:
Inclusion Criteria:

* case reported in the World Health Organization (WHO) database of individual safety case report to 11/20/2018
* Patient treated with at least one bDMARD prescriptions
* adverse events reported were including the MedDRA terms

Exclusion Criteria:

* Chronology not compatible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with one bDMARD
Sampling Method: Non-Probability Sample
Enrollment: 594226 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-06-28 (Estimated); Study Completion 2019-06-28 (Estimated)

PRIMARY OUTCOMES:
Risk of reporting cancer overall specific cancers | Reported in the World Health Organization (WHO) database of individual safety case reports to 12/31/2018
  Estimate statistically the risk of reporting cancer overall and specific cancers (including breast, lung, lymphoma, cervical, melanoma and NMSC) compared with all other adverse drug reactions (ADR) for abatacept compared to all ADRs for other bDMARDs performing a disproportionality analysis
Risk of reporting specific cancers | Reported in the World Health Organization (WHO) database of individual safety case reports to 12/31/2018
  Estimate statistically the risk of specific cancers (including breast, lung, lymphoma, cervical, melanoma and NMSC) compared with all other adverse drug reactions (ADR) for abatacept compared to all ADRs for other bDMARDs performing a disproportionality analysis

CONTACTS AND LOCATIONS:
Overall Officials: François MONTASTRUC, PhD MD, Study Director — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

REFERENCES:
- [Derived] de Germay S, Bagheri H, Despas F, Rousseau V, Montastruc F. Abatacept in rheumatoid arthritis and the risk of cancer: a world observational post-marketing study. Rheumatology (Oxford). 2020 Sep 1;59(9):2360-2367. doi: 10.1093/rheumatology/kez604. PMID 31880308